CLINICAL TRIAL: NCT03950986
Title: Increasing Vaccine Uptake Among Veterans at the Atlanta VA Health Care System Through a Randomized Trial
Brief Title: Increasing Vaccine Uptake Among Veterans at the Atlanta VA Health Care System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Atlanta VA Medical Center (U.S. Federal Agency)
Collaborators: General Services Administration (GSA) (U.S. Federal Agency); Emory University (Other)
Responsible Party: Principal Investigator, Vincent Marconi, Director of Infectious Diseases Research, Atlanta VA Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AtlantaVAMC
Record Dates: First submitted 2019-04-25; First posted 2019-05-15 (Actual); Last update posted 2020-01-10 (Actual); Status verified 2020-01

CONDITIONS: Influenza; Tetanus; Diphtheria; Pertussis; Pneumonia
Keywords: Vaccination; EHR Reminders; Nudge; Electronic Medical Records; Behavioral Economics
MeSH Terms: conditions — Influenza, Human; Tetanus; Diphtheria; Whooping Cough; Pneumonia

STUDY DESIGN:
Intervention Model Description: Intervention is designed to target patients of primary care providers (physicians, physician assistants and nurse practitioners) in the Atlanta VA Medical System. Primary care providers will be assigned to a provider-side treatment (modified vaccine reminders in the electronic health record (EHR) system) or to control (existing vaccine reminders). Outcomes will be tracked for patients who have appointments with these providers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Providers assigned to the control group will receive unmodified vaccine reminders (as they already appear in the VA EHR system). Separate reminders will appear for the different vaccines of interest.
- Treatment (Experimental): Providers in the treatment group will receive modified clinical reminders for the vaccines of interest. Reminders for the different vaccines of interest will be bundled into a single reminder, and other changes made to streamline the design and reduce provider burden. Other changes include an immunization dashboard that relays a patient's vaccination status and talking points for providers to use in their dialogues with patients.
  Interventions: Other: Modified clinical reminders

INTERVENTIONS:
Other: Modified clinical reminders — Clinical reminders for the vaccines of interest will be bundled into a single reminder, and other changes made to streamline the design and reduce provider burden. Other changes include an immunization dashboard that relays a patient's vaccination status and talking points for providers to use in their dialogues with patients.
  Arms: Treatment

SUMMARY:
The Office of Evaluation Sciences is collaborating with Emory University and the Atlanta VA Health Care System to increase adult immunizations uptake among veterans. The intervention targets patients of primary care providers (physicians, physician assistants and nurse practitioners) through a modification of the existing reminders in the VA electronic health record system. The team will evaluate the intervention using a randomized controlled trial.

DETAILED DESCRIPTION:
The Office of Evaluation Sciences is collaborating with Emory University and the Atlanta VA Health Care System to increase adult immunizations uptake among veterans. The intervention targets patients of primary care providers (physicians, physician assistants and nurse practitioners) through a modification of the existing reminders in the VA electronic health record system.

The intervention includes a bundled vaccination reminder for influenza, pneumococcal and TDap vaccines, an immunization dashboard that relays a patient's vaccination status and history, and talking points for providers to use in their dialogues with patients. This intervention was designed to mitigate potential bottlenecks to vaccination, based on conversations and observations with facility clinicians.

The team will evaluate the intervention using a randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* All patients must have appointments with active primary care providers (physicians, physician assistants and nurse practitioners) in the Atlanta VA Health Care System

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 67000 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Percent of patients receiving one of more vaccines of interest when due for these vaccines | 6 months
  Percent of patients receiving of one or more of the influenza, pneumococcal (PCV13 or PPSV23) or Tdap/Td vaccines during the observation period, conditional on the patient being due for at least one of these vaccines at any appointment during the observation period
Percent of patients receiving the influenza vaccine when due for the vaccine | 6 months
  Percent of patients receiving the influenza vaccine during the observation period, conditional on the patient being due for the influenza vaccine at any appointment during the observation period

SECONDARY OUTCOMES:
Percent of patients receiving Tdap/Td or pneumococcal vaccines when due | 6 months
  Percent of patients receiving Tdap/Td or pneumococcal vaccines during the observation period, conditional on the patient being due for at least one of these vaccines at any appointment during the observation period
Cost per additional individual vaccinated | 6 months
  Should these data be available, will assess the cost per additional individual vaccinated

CONTACTS AND LOCATIONS:
Overall Officials: Pompa Debroy, MS, Principal Investigator — Office of Evaluation Sciences, U.S. General Services Administration; Russ Burnett, PhD, Principal Investigator — Office of Evaluation Sciences, U.S. General Services Administration; Saad Omer, MBBS, MPH, PhD, Principal Investigator — Emory University; Joseph M Wallace, Principal Investigator — Atlanta VA Health Care System; Vincent Marconi, MD, Principal Investigator — Atlanta VA Health Care System, Emory University
Locations (1):
- Atlanta VA Medical Center, Decatur, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Debroy P, Balu R, Burnett R, Johnson RA, Kappes HB, Wallace JM, Marconi VC. A cluster randomized controlled trial of a modified vaccination clinical reminder for primary care providers. Health Psychol. 2023 Mar;42(3):195-204. doi: 10.1037/hea0001218. Epub 2022 Oct 13. PMID 36227309
- See also: Project Analysis Plan — https://oes.gsa.gov/projects/increasing-adult-vaccines-atlanta-va/

DOCUMENTS (1):
  • Statistical Analysis Plan (2019-04-17): https://cdn.clinicaltrials.gov/large-docs/86/NCT03950986/SAP_000.pdf